CLINICAL TRIAL: NCT07234487
Title: Randomized Study Comparing AVD Combined With Fixed-Dose Nivolumab Versus PET-Adapted BEACOPP-like Regimen as First-Line Treatment in Advanced Classical Hodgkin Lymphoma
Brief Title: Comparison of AVD + Low-Dose Nivolumab vs. PET-Adapted BEACOPP-like in Advanced cHL
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: St. Petersburg State Pavlov Medical University (Other)
Responsible Party: Principal Investigator, Ivan S Moiseev, Vice-director of RM Gorbacheva Research Institute, St. Petersburg State Pavlov Medical University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 28/24-н
Record Dates: First submitted 2025-02-03; First posted 2025-11-18 (Actual); Last update posted 2025-11-18 (Actual); Status verified 2025-04

CONDITIONS: Hodgkin Lymphoma
Keywords: Hodgkin Lymphoma; N-AVD; nuvolumab; BEACOPPesc; Low dose nivolumab
MeSH Terms: conditions — Hodgkin Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Nivo-AVD (Experimental): Nivo-AVD cohort patients will receive 2 cycles of nivolumab monotherapy (40 mg) followed by Nivo-AVD combination therapy (6 cycles total)
  Interventions: Drug: Nivo-AVD
- BEACOPP-like regimes - Standard cohort (Active Comparator): In the Standard cohort, patients will receive therapy according to current clinical guidelines for first-line therapy of cHL, which include starting first-line therapy with 2 cycles of BEACOPP-like regimens and, after assessing response after 2 courses, switching to an A(B)VD regimen (when achieving CR by PET/CT) or continuing therapy with BEACOPP-like regimens (when achieving PR,SD by PET/CT)
  Interventions: Drug: BEACOPP-like

INTERVENTIONS:
Drug: Nivo-AVD — 1. Monotherapy phase - Nivolumab - 40 mg every 14 days x 2 cycles
  2. Combination therapy phase - Nivo-AVD x 6 cycles Nivolumab - 40 mg every 14 days; Doxorubicin 25 mg/m2 in D1 and 15; Vinblastine 6 mg/m2 (no more than 10 mg) in D 1 and 15; Dacarbazine 375 mg/m2 in D 1 and 15;
  Arms: Nivo-AVD
Drug: BEACOPP-like — * BEACOPP-like regimens x 2 cycles + BEACOPP-like regimens x 4 (for patients with PR, SD by PET/CT after 2 cycles)
  * BEACOPP-like regimens x 2 + A(B)VD x 4 cycles (for patients with CR by PET/CT after 2 cycles)
  Arms: BEACOPP-like regimes - Standard cohort

SUMMARY:
Patients in this prospective multicenter phase II study will be randomized between two first-line therapy strategies for advanced stages of cHL. In the Nivo-AVD cohort, patients will receive 2 cycles of nivolumab monotherapy followed by a switch to Nivo-AVD combination therapy (total of 6 cycles); in the Standard cohort, patients will receive therapy according to current clinical guidelines in Russian Federation for first-line therapy of cHL, which include starting first-line therapy with 2 cycles of BEACOPP-like regimens and, after assessing response after 2 courses, switching to A(B)VD or continuing with BEACOPP-like regimens

ELIGIBILITY:
Inclusion Criteria:

* Patients with newly diagnosed histologically confirmed stage IIB, III or IV classical hodgkin lymphoma who have not previously received specific therapy;
* Patients with evidence of lesion extent assessed by whole-body PET/CT;
* Patients aged 18-60 years;
* ECOG 0-2;
* Use of highly effective contraceptive methods from the moment of signing the informed consent form, throughout the study and within 6 months after receiving the last dose of the drug;

Exclusion Criteria:

* Severe organ failure: creatinine > 2 norms; alanine aminotransferase, aspartate aminotransferase > 5 norms; bilirubin> 1.5 norms;
* Respiratory failure > grade 1 at the time of enrollment
* Requirement for vasopressor support at the time of enrollment
* Uncontrolled bacterial or fungal infection at the time of enrollment
* Active or prior documented autoimmune disease requiring systemic treatment
* Pregnancy, breastfeeding, planning pregnancy or parenthood during the study period
* Hypersensitivity or allergy to study drugs
* Somatic or mental pathology that does not allow to perform research procedures, including the signing of informed consent
* Simultaneous use of drugs or medical devices studied in other clinical trials

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 178 (Estimated)
Dates: Start 2024-10-14 (Actual); Primary Completion 2029-10 (Estimated); Study Completion 2030-10 (Estimated)

PRIMARY OUTCOMES:
Incidence of adverse events | Up to 24 months from thetreatment start
  To compare the safety of therapy use in the Nivo-AVD and Standard cohorts: analysis of the incidence, severity and spectrum of adverse events (according to CTCAE v5.0 criteria)

SECONDARY OUTCOMES:
Progression-free survival | 12, 24 and 36 months after completion of therapy
  To compare progression-free survival in the Nivo-AVD and Standard cohorts
Response rates | after 2 cycles of nivo and 2 cycles of Nivo-AVD (3 months from therapy initiation) and at the end of treatment (7 months from therapy initiation) and, in Standard cohorts, after 2 cycles and EOT of BEACOPPesc (2 and 6 months)
  To compare the rates of objective response, complete and partial responses after 2 and 6 courses of therapy in the Nivo-AVD and Standard cohorts by whole-body PET-CT (according to Lugano criteria for chemotherapy and LYRIC criteria for immunochemotherapy)
Overall survival | 12, 24, and 36 months after completion of therapy
  - To compare overall survival at 12, 24, and 36 months after completion of therapy in the Nivo-AVD and Standard cohorts.

CONTACTS AND LOCATIONS:
Overall Officials: Natalia Mikhailova, MD, PhD, Study Chair — St. Petersburg State Pavlov Medical University
Locations (1):
- St. Petersburg State Pavlov Medical University, Saint Petersburg, Russia